CLINICAL TRIAL: NCT07156084
Title: Persistence of Immune Response Six Years After One Dose of 9vHPV Vaccine Among Male and Female Students
Acronym: CIRN-HPV-ONE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Canadian Immunization Research Network (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CT-26 CIRN HPV 1 dose
Record Dates: First submitted 2025-08-02; First posted 2025-09-04 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: HPV Vaccine
Keywords: HPV; Vaccination; Schedule

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- One HPV vaccine dose received 6 years before recruitment (Experimental)
  Interventions: Biological: HPV nonavalent vaccine (Gardasil-9)

INTERVENTIONS:
Biological: HPV nonavalent vaccine (Gardasil-9) — One dose HPV nonavalent vaccine

SUMMARY:
Since the 2019-2020 school year, the province of Quebec (Canada) has been administering one dose of nonavalent (9vHPV) vaccine to students of all genders in Grade 4 of elementary school through the school-based program.

Little data on the immunogenicity (antibody production) and long-term efficacy of a single dose of the vaccine are available, particularly in boys.

The primary objective of this study is to assess the persistence of HPV antibodies six years after the administration of a single dose of the 9vHPV vaccine to students aged 9 to 11 years in Grade 4 in 2019-2020.

The study will be conducted at the CHU de Québec-Université Laval research center.

Recruitment is conducted through school service centers in the Quebec City region. Youth who received only a single dose of the 9vHPV vaccine at the ages of 9-11 in 2019-2020 will be eligible to participate.

Approximately 300 youth will take part in this study: 150 girls and 150 boys.

Participants will have to answer few questions about their health to ensure their eligibility for the study. For eligible participants consenting to participate a 10 ml (<1 tablespoon) blood sample will be taken.

DETAILED DESCRIPTION:
Since the 2019-2020 school year, the province of Quebec (Canada) has been administering one dose of nonavalent (9vHPV) vaccine to students of all genders in Grade 4 of elementary school through the school-based program. The second dose, which was to be administered five years after the first, was never administered following a recommendation from the Quebec Committee (of Experts) on Immunization (CIQ) in 2024. The current recommendation is to administer a single dose of 9vHPV vaccine to all immunocompetent individuals aged 9 to 20 years. The Canadian expert committee (National Advisory Committee on Immunization) and the World Health Organization (WHO) expert committee have made the same recommendation.

Little data on the immunogenicity (antibody production) and long-term efficacy of a single dose of the vaccine are available, particularly in boys.

The results of this study will allow for a better assessment of the immunity provided by a single dose of the HPV vaccine at the time when young people begin their sexual life and are exposed to HPV.

The primary objective of this study is to assess the persistence of HPV antibodies six years after the administration of a single dose of the 9vHPV vaccine to students aged 9 to 11 years in Grade 4 in 2019-2020.

The study will be conducted at the CHU de Québec-Université Laval research center, in the Vaccination Research Team clinic located in Quebec City.

Recruitment is conducted through school service centers in the Quebec City region. Youth who received only a single dose of the 9vHPV vaccine at the ages of 9-11 in 2019-2020 will be eligible to participate.

Approximately 300 youth will take part in this study: 150 girls and 150 boys.

Participants will have to answer few questions about their health to ensure their eligibility for the study. For eligible participants consenting to participate a 10 ml (<1 tablespoon) blood sample will be taken.

ELIGIBILITY:
Inclusion Criteria:

* Have received a single dose of 9vHPV vaccine at ages 9-11 during the school year 2019-2020;
* Not have received any other HPV vaccine doses;
* Be able to consent to the study.

Exclusion Criteria:

* Immunosuppressed (at recruitment or when immunized).

Ages: 15 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2025-09-23 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Detectable antibodies | At recruitment (6 years post-one HPV vaccine dose)
  Proportion of participants with detectable antibodies
Geometric mean concentrations | At recruitment (6 years post-one HPV vaccine dose)
  Geometric mean concentrations of antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Chantal Sauvageau, MD, Principal Investigator — INSPQ and Laval University
Locations (1):
- Centre de recherche du CHU de Québec-Université Laval, Québec, Quebec, Canada